CLINICAL TRIAL: NCT05577221
Title: Effect of High Flow Nasal Air on Dyspnea During Weaning From Mechanical Ventilation
Brief Title: High Flow During Weaning From Mechanical Ventilation
Acronym: FLOWEAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP221010
Record Dates: First submitted 2022-09-26; First posted 2022-10-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Acute Respiratory Failure
Keywords: Dyspnea; Weaning; Mechanical ventilation; High flow nasal air
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Collection of physiological parameters (Experimental): Installation of the high-flow humidified nasal oxygen therapy device and variation of the inspiratory flow rate (0 L/min, 30 L/min, 50 L/min and 70 L/min) then the weaning test will be performed. During each step of the protocol (= each variation of the inspiratory flow), the intensity of dyspnea will be collected, the esophageal pressure will be measured, the respiratory drive (P0.1) will be measured, the EMG of the respiratory muscles will be measured and the comfort will be measured. Each step lasts about 15 minutes with 5 minutes of wash-out before the next step. Once the 4 steps will be conducted, the weaning test will be performed (without wash-out), for a duration of one hour, 30 minutes with high flow humidified nasal oxygen (50 L/min) and 30 minutes without (both steps being randomized. The whole protocol will last 2h15.
  Interventions: Device: High Flow Nasal Air

INTERVENTIONS:
Device: High Flow Nasal Air — Administration of air at high flow by using a high flow nasal oxygenation (FiO2 21%) device
  Other Names: High Flow Nasal Cannula

SUMMARY:
Detection and relief of dyspnea in mechanically ventilated patients is a priority. Optimization of mechanical ventilation settings is unfortunately often insufficient to relieve dyspnea in patients entering the weaning process. Pharmacological treatments are effective but their use is likely to delay separation with the ventilator. Promoting the development of non-pharmacological interventions is therefore an interesting avenue. The hypothesis is that the application of high-flow humidified nasal air in orotracheally intubated patients can decrease the work of breathing and relieve dyspnea at the time of weaning from mechanical ventilation. Patients will be exposed to stepwise increase in high flow nasal air (0 L/min, 30 L/min, 50 L/min and 70 L/min) before to undergo a 60 minutes spontaneous breathing trial. During the protocol, dyspnea, inspiratory effort, respiratory drive, respiratory muscles electromyogram (EMG) and patient's comfort will be assessed.

DETAILED DESCRIPTION:
Patients equipped with an esophageal probe and deemed ready to undergo a spontaneous breathing trial will be included.

During, the inclusion visit, main characteristics of the patients and ICU stay will be collected in the patient's chart: age, sex, comorbidities, date of admission to intensive care, date of intubation, severity score (SOFA), reason for admission to intensive care , weight, height, ventilation settings, P0.1, respiratory rate, SpO2, dyspnea and comfort score.

Secondarily, the quality of the esophageal pressure signal will be checked. Esophageal pressure will be collected using a nasogastric tube (NutriventTM, SIDAM, Italy). Esophageal pressure will be measured continuously by the Labchart system installed on the department's dedicated computer.

Third, the EMG collection device will be implemented. EMG signals will be collected by surface electrodes on the scalene and intercostal muscles and on the sides of the nose. The electrodes are connected to collection modules operating with the LabChart system.

Finally, the high-flow humidified air device will be installed (AIRVO 2; Fisher and Paykel Healthcare, Auckland, New Zealand) and nasal cannulas adapted to the patient's anatomy will be positioned. The FiO2 will be fixed at 21% for the duration of the study. The flow will be set at 0 L/min at the inclusion visit. The humidified air temperature will be set to 37°C.

The protocol will consist of installing the high-flow humidified nasal oxygen therapy device and varying the nasal flow (4 different conditions: 0 L/min, 30 L/min, 50 L/min and 70 L/min) then performing the spontaneous breathing trial (duration 60 minutes). During each of the steps of the protocol, a collection of the intensity of the dyspnea, a measurement of the esophageal pressure, a measurement of the respiratory drive, an EMG measurement of the respiratory muscles and a comfort assessment will be carried out.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. orotracheal intubation
3. Decision to initiate a spontaneous breathing trial by the clinical team
4. Visual analogic scale of dyspnea > 3/10
5. Informed consent to participate
6. Patient covered by the national health

Exclusion Criteria:

1. No esophageal probe in place
2. Extubation planned without a spontaneous breathing trial
3. Glasgow coma scale< 12
4. Patient's refusal
5. No coverage by the national health insurance
6. Patient under legal protection of justice

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-02-17 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
The effect of high-flow humidified nasal oxygen therapy on dyspnea in orotracheally intubated patients at the time of weaning from mechanical ventilation. | at inclusion, compare to 15, 35, 55, 75, 105 and 135 min
  Dyspnea Numerical Rating Scale from 0 to 10
The effect of high-flow humidified nasal oxygen therapy on dyspnea in orotracheally intubated patients at the time of weaning from mechanical ventilation. | at inclusion, compare to 15, 35, 55, 75, 105 and 135 min
  Mechanical Ventilation Respiratory Distress Observational Scale

SECONDARY OUTCOMES:
inspiratory effort | at inclusion, compare to 15, 35, 55, 75, 105 and 135 min
  Amplitude of the esophagus pressure
respiratory drive | at inclusion, compare to 15, 35, 55, 75, 105 and 135 min
  inspiratory occlusion pressure (P0.1)
respiratory muscles activity | at 15 min to inclusion, compare to, 35, 55, 75, 105 and 135 min
  electromyogram of the respiratory muscles
patient comfort | at inclusion, compare to 15, 35, 55, 75, 105 and 135 min
  Visual analogic scale. Scale of 1 to 10 with 10 corresponding to minimal comfort

CONTACTS AND LOCATIONS:
Locations (1):
- Medical ICU R3S, Pitié-Salpétriêre Hospital, Paris, France